CLINICAL TRIAL: NCT01738906
Title: The Effect of Moderate Alcohol Consumption on Subsequent Food Reward
Brief Title: The Effect of Alcohol on Food Reward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henk FJ Hendriks (Other)
Collaborators: Foundation for Alcohol Research (SAR), The Netherlands (Unknown); Ministry of Economic Affairs, The Netherlands (Unknown)
Responsible Party: Sponsor-Investigator, Henk FJ Hendriks, Project Manager, TNO
Organization: TNO (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: P9532
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Body Weight
MeSH Terms: conditions — Obesity; Body Weight | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Alcohol placebo and MSF (Experimental): 175 mL orange juice with 31 g Fantomalt maltodextrin and modified sham feeding of 40 g butter cake
  Interventions: Other: Orange juice; Other: maltodextrin; Other: butter cake MSF
- Alcohol and MSF (Experimental): 65 mL vodka with 135 mL orange juice (ca 20 g alcohol)and modified sham feeding of 40 g butter cake
  Interventions: Other: Orange juice; Other: Vodka; Other: butter cake MSF
- Alcohol placebo and consumption (Experimental): 175 mL orange juice with 31 g maltodextrin and consumption of 40 g butter cake
  Interventions: Other: Orange juice; Other: maltodextrin; Other: butter cake consumption
- Alcohol and consumption (Experimental): 65 mL vodka with 135 mL orange juice and consumption of 40 g butter cake
  Interventions: Other: Orange juice; Other: Vodka; Other: butter cake consumption
- Alcohol placebo and control (Experimental): 175 mL orange juice with 31 g maltodextrin and no oral exposure to butter cake
  Interventions: Other: Orange juice; Other: maltodextrin
- Alcohol and control (Experimental): 65 mL vodka with 135 mL orange juice and no oral exposure to butter cake
  Interventions: Other: Orange juice; Other: Vodka

INTERVENTIONS:
Other: Orange juice
  Other Names: Orange Juice (Appelsientje)
Other: maltodextrin
  Other Names: Fantomalt maltodextrin (energy powder), Nutricia
  Arms: Alcohol placebo and MSF; Alcohol placebo and consumption; Alcohol placebo and control
Other: Vodka
  Other Names: Smirnoff Vodka
  Arms: Alcohol and MSF; Alcohol and consumption; Alcohol and control
Other: butter cake MSF — chewing on 40 gram cake for 6 minutes and before swallowing expectorating the bolus in cup.
  Other Names: cake modified sham feeding
  Arms: Alcohol and MSF; Alcohol placebo and MSF
Other: butter cake consumption — chewing for 6 min on 40 gram cake and then swallow it.
  Other Names: cake consumption
  Arms: Alcohol and consumption; Alcohol placebo and consumption

SUMMARY:
Rationale

It has been shown in several studies that alcohol increases subsequent food intake. However, moderate alcohol consumption has no clear effects on hunger and satiety hormones. In the Western world, where palatable food is highly available, food reward may play an important role in food intake. Alcohol consumption is known to stimulate neurotransmitters important for food reward and may therefore stimulate the reward response on a subsequent meal. This may lead to higher food consumption than when no alcohol is consumed. It is hypothesized that the reward response of food or beverages can already be generated when food or beverages are sensed in the mouth, because oral nutrient sensing is known to induce a satiety response (i.e. the cephalic phase response). Moreover, taste buds directly signal brain areas closely connected to the reward areas in the brain.

Primary objective

* To determine whether moderate alcohol consumption influences subsequent food reward, as measured by questionnaires on food 'wanting' and food 'liking', and salivary and blood parameters related to reward.

Secondary objectives

* To determine whether food reward is different when food is consumed than when food is sensed in the mouth, as measured by questionnaires on food 'wanting' and food 'liking', and salivary and blood parameters related to food reward.
* To determine whether moderate alcohol consumption influences subsequent food reward differently when food is consumed than when food is sensed in the mouth, as measured by questionnaires on food 'wanting' and food 'liking', and salivary and blood parameters related to food reward.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men;
* Age 25-50 years on the day of the screening;
* Body Mass Index (BMI) of 20-25 kg/m2;
* Body weight of 60-100 kg;
* Able to read, write and fully understand the Dutch language, and
* Able to participate int he sudy, willing to give written informed consent and to comply with the study procedures and restrictions.

Exclusion Criteria:

* Above average score (>2.26) on the restrained scale of the Dutch Eating Behaviour Questionnaire;
* Alcohol consumption <6 and >20 standard glasses/week;
* Not having regular and normal Dutch eating habits;
* Not having a normal day/night rhythm;
* Smoking, or stopped with smoking <3 months prior to start of the study;
* Using drugs, or stopped using drugs <3 months prior to start of the study;
* Having a (family) history of alcohol or drug related problems;
* Reported slimming or being on a medically described diet;
* Having a vegan, vegetarian or macrobiotic lifestyle;
* Loss of blood outside the limits of Sanquin within 3 months prior to screening;
* Participation in a clinical trial within 3 months prior to the start of this study or more than 4 times a year;
* Having a food allergy, sensitivity or disliking one of the foods used in the study;
* Reported unexplained weight loss or gain of >4 kg in the month prior to the screening;
* Inappropriate veins for cannula insertion;
* Not having a general practitioner or health insurance;
* Having a history of medical or surgical events or disease that may significantly affect the study outcome, particularly physiological disorders, metabolic or endocrine disease and gastrointestinal disorders; and/or
* Any condition which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol.

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Explicit food 'wanting' | up to 75 minutes
  Questionnaire measuring food 'wanting' explicitly with the question: "How much do you want to eat at this moment?" This is scored on a visual analogue scale ranging from 0-100.
Implicit food 'wanting' for different food categories | up to 30 minutes
  Computer task measuring food 'wanting' implicitly for different food categories. This is a forced choice task in which subjects have to choose as quick and precise the food product they want to eat most at that moment.
explicit food 'wanting' for different food categories | up to 30 minutes
  Questionnaire measuring food wanting explicitly for different food categories on a visual analogue scale (ranging 0-100).
explicit food 'liking' for different food categories | up to 30 minutes
  Questionnaire measuring food 'liking' for different food categories on a visual analogue scale (ranging 0-100).

CONTACTS AND LOCATIONS:
Overall Officials: Henk Hendriks, PhD, Principal Investigator — TNO Zeist, The Netherlands
Locations (1):
- Centre for Human Drug Research (CHDR), Leiden, South Holland, Netherlands